CLINICAL TRIAL: NCT02565823
Title: Investigation of Exercise-Induced Myokines and Adipokines
Brief Title: The Effects of Exercise of Secreted Factors From Muscle and Adipose Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Principal Investigator, Laurie Goodyear, PhD, Joslin Diabetes Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHS2015-11
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise intervention (Experimental): Subjects will undergo an acute bout of exercise for 45 mins at 75% of peak aerobic capacity
  Interventions: Other: Exercise bout

INTERVENTIONS:
Other: Exercise bout — Participants will exercise for 45min at 75% of VO2peak

SUMMARY:
The purpose of this study is to find out whether exercise leads to changes in the blood that are produced by exercised muscles and if these changes produce new hormones that affect the body's regulation of sugar and body weight.

DETAILED DESCRIPTION:
Recent work in the laboratory at the Joslin Diabetes Center and elsewhere has shown that when small animals exercise they improve their muscles and improve their blood sugar levels. Also, these animals show changes in their abdominal fat tissue, compared to animals that did not exercise. Our data suggest that factors released from exercised muscle and fat tissue from exercised mice also has a positive effect on other tissues in the same animal. Therefore, there could be new factors or hormones, which come from the trained animals' muscles or fat tissue and which exert a positive effect on the animals' blood sugar levels. Large studies with human volunteers have shown that exercise can improve blood sugar uptake into skeletal muscle and lower blood sugar levels, thereby preventing type 2 diabetes. The purpose if this study is to evaluate if a single exercise bout leads to changes in circulating factors in the blood. We plan to detect if there are hormones being produced in the body that have a beneficial effect elsewhere in the body.

ELIGIBILITY:
Inclusion Criteria:

- Age between 18-35. Body mass index (BMI) must be ≥20 and ≤26 kg/m2. HbA1c values ≤5.7%

Exclusion Criteria:

- Age <18 and >35; HbA1c ≥ 5.7%; heart or lung disease; acute systemic infection accompanied by fever, body aches, or swollen lymph glands; BMI ≥ 26 kg/m2; current dieting or weight loss efforts; current pregnancy or breastfeeding; known history of HIV/AIDS; cancer; biochemical evidence of renal or hepatic dysfunction; renal or liver disease; demyelinating diseases such as multiple sclerosis or amyotrophic lateral sclerosis; recent blood donation; clinical history of stroke; hypertension (systolic > 140 mmHg or diastolic > 90 mmHg); type 1 or 2 diabetes; history of keloid formation inability to exercise at 50% of predicted heart rate (HR) reserve at baseline. Participants taking beta-blockers Participants who screen positive for The American Heart Association's contraindications to exercise testing

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in myokines/adipokine concentration | baseline, and 15, 45 and 1h:45 mins after exercise session.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie J. Goodyear, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States